CLINICAL TRIAL: NCT01884038
Title: A Single Center, Randomized, Double-Blind, Parallel Placebo-Controlled Study of the Safety and Efficacy of Perioperative Remodulin® in Orthotopic Liver Transplant Recipients
Brief Title: Safety and Efficacy of Perioperative Remodulin® in Orthotopic Liver Transplant Recipients
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RIV-LT-301
Record Dates: First submitted 2012-10-19; First posted 2013-06-21 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2013-06

CONDITIONS: Liver Transplant
Keywords: Liver Transplant; Prostacyclin; Treprostinil sodium; Remodulin; Reperfusion Injury; Primary Nonfunction
MeSH Terms: conditions — Reperfusion Injury | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remodulin (Experimental): Remodulin initiated as a continuous IV infusion at a dose of 2.5 ng/kg/min after subjects have been assessed as hemodynamically stable in the ICU. Dose may be escalated in 1.25- to 2.5-ng/kg/min increments, up to 7.5 ng/kg/min, with a target dose of 5 ng/kg/min, based on tolerability. The dose will be maintained at the maximum tolerated dose, not to exceed 7.5 ng/kg/min for 5 days after the transplantation surgery.
  Interventions: Drug: treprostinil sodium
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: treprostinil sodium — A single dose strength of treprostinil sodium (1.0 mg/mL) and matching placebo will be provided in 20-mL multi-dose vials.
  The study drug will be started after induction of anesthesia and increased incrementally to a target dose of 10 ng/kg/min during surgery and 48 hours post-operative
  Other Names: Remodulin; UT 15
  Arms: Remodulin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Patients undergoing orthotopic liver transplant will experience some degree of clinical and/or biochemical hepatic dysfunction. This early injury is known as primary graft dysfunction and varies from minor abnormalities to primary nonfunction. Prostaglandin-class drugs, including prostacyclin and its analogs, could represent an important advance toward the goal of reducing transplant related morbidity, mortality and associated costs by providing these benefits.

DETAILED DESCRIPTION:
In vitro and in vivo research has consistently demonstrated an array of potential beneficial effects of prostanoids under both immune and non-immune circumstances relevant to liver allografts. (1-3) Recent reviews summarize the pharmacologic rationale and nonclinical and clinical experience supporting for the use of prostanoids, including prostacyclin and its analogs, in reducing early morbidity and mortality associated with liver transplantation. Prostaglandin-class drugs, including prostacyclin and its analogs, could represent an important advance toward the goal of reducing transplant related morbidity, mortality and associated costs by providing these benefits. Additionally, the reduction in serum creatinine and reduced need for post-operative dialysis observed in some studies has implications in protecting the kidneys from the nephrotoxic affects of the immunosuppressant agents, especially during the early post-operative period.

As a chemically stable analog of prostacyclin (PGI2), peri-operative intravenous administration of Remodulin is hypothesized to ameliorate or prevent reperfusion damage and thereby decrease hospitalization time and improve the clinical outcome of liver transplantation, compared to placebo control. Remodulin, as a prostanoid, is expected to facilitate restoration of the blood supply to the revascularized graft, and to provide the well-characterized protective effects of this class of compounds in liver transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Accepted as a liver transplant candidate at the University of Pittsburgh Medical Center
* Be receiving a cadaver donor liver transplant
* Treated in accordance with the standard of care protocol(s) in effect for liver transplant recipients at the University of Pittsburgh Medical Center.

Exclusion Criteria:

* Receiving a living done liver transplant
* Receiving a donor liver with a cold ischemia time less that 6 hours
* Receiving a donor liver with macrosteatosis greater than 30%
* Receiving any investigation drug with the except of alemtuzamab (Camphath)
* Failed liver transplant in previous 180 days
* Prior organ transplant or cell infusion
* Undergoing multi-organ transplant
* Pregnant or nursing female

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Duration of the initial hospitalization (days) following transplantation | up to 180 days
Area under the curve (AUC) of serum aspartate transaminase (AST) levels. | 7 days
  The difference in serum AST as measured by AUC during the first seven days post-transplant will be compared between placebo and Remodulin treatment groups. AST is a serum transaminase marker of hepatic injury, and the AUC of AST levels represents the total magnitude of injury the liver experiences against time.

SECONDARY OUTCOMES:
Serum AST and alanine transaminase (ALT ) levels after transplant (Peak and Area Under the Curve [AUC]) | 7 days
Primary allograft nonfunction defined as patient death or retransplant within 30 days due to liver failure | 30 days
Graft survival | 30 days, 90 days and 180 days
Subject survival at | Day 30, 90, and 180
Post-transplant renal function | 30 days
Duration of time spent in the intensive care unit (ICU; days) during the initial hospitalization. | up to 180 days
Intra-operative blood product usage | 1 day
Death from any cause | 180 days
Total costs for initial transplant hospitalization | up to 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Amadeo Marcos, MD, Principal Investigator — University of Pittsburgh Medical Center; Raman Venkataramanan, Ph.D, F.C.P., Principal Investigator — University of Pittsburgh Medcial Center
Locations (1):
- University of Pittsburgh Medical Center, Starzl Transplantation Institute, Pittsburgh, Pennsylvania, United States